CLINICAL TRIAL: NCT06391723
Title: Clinical, Cognitive and Neural Effect of Potentiation of Electroconvulsive Therapy (ECT) by Repetitive Transcranial Magnetic Stimulation (rTMS) at 10 ECT in Patients With Characterized Pharmacoresistant Depressive Episode
Brief Title: Clinical, Cognitive and Neural Effects of Potentiation of ECT by rTMS in Treatment-Resistant Depression
Acronym: STIMAGNECT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Rouvray (Other Government)
Collaborators: University Hospital, Rouen (Other); Centre Hospitalier Sainte Anne, Paris (Unknown)
Responsible Party: Principal Investigator, Maud Rothärmel, Principal investigator, Centre Hospitalier du Rouvray
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-A01813-42
Record Dates: First submitted 2024-01-30; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
Keywords: Treatment-resistant-depression; repetitive transcranial magnetic stimulation (rTMS); electroconvulsive therapy (ECT); combination of neurostimulation techniques
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, sham-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS group (Active Comparator): 5 active rTMS before starting ECT, then from the sixth ECT session, an active rTMS session will occur the day before each ECT session
  Interventions: Device: Active rTMS
- Sham rTMS group (Placebo Comparator): 5 sham rTMS before starting ECT, then from the sixth ECT session, a sham rTMS session will occur the day before each ECT session
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — rTMS will be administered over the left dorsolateral prefrontal cortex (20 Hz, 90% resting motor threshold, 20 2 s trains with 60-s intervals, 800 pulses/session)
  Arms: Active rTMS group
Device: Sham rTMS — Sham rTMS will be administered over the left dorsolateral prefrontal cortex
  Arms: Sham rTMS group

SUMMARY:
Electroconvulsive therapy (ECT) is one of the most effective treatments for treatment-resistant depression (TRD). However, due to response delay and cognitive impairment, ECT remains an imperfect treatment. In this multicenter, randomized, double-blind, sham-controlled study, our objective is to assess the priming effect of rTMS sessions before ECT on clinical, cognitive and neural response in patients with TRD.

DETAILED DESCRIPTION:
80 patients with TRD will be assigned to active or sham rTMS before ECT treatment. Five sessions of active/sham rTMS will be administered over the left dorsolateral prefrontal cortex (20 Hz, 90% resting motor threshold, 20 2 s trains with 60-s intervals, 800 pulses/session) before ECT (which was active for all patients) started. Then, from the sixth ECT session, an rTMS session will occur the day before each ECT session. Clinical assessment, cognitive assessment and brain imaging (structural MRI, resting state functional MRI, MR spectroscopy) will take place before and after 10 ECT sessions. Clinical, cognitive and neural changes will be compared between both groups after 10 ECT sessions.

The primary outcome will be the response rate after 10 ECT, i.e. the percentage of patients who achieved a reduction of 50% or more from their initial Hamilton Depression Scale score (HAMD-21 items).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Major Depressive Disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria
* HAMD score ≥15
* In case of unipolar disorder: no remission after at least two different antidepressants prescribed at a dose and duration sufficient for the current episode
* In the case of bipolar disorder: no remission despite lithium at an adequate plasma level combined with lamotrigine or quetiapine monotherapy at full dose
* No change of antidepressant or mood stabilizer treatment for at least 15 days
* To be rTMS-naive
* Without benzodiazepine or antiepileptic treatment for at least 15 days
* To understand spoken and written French
* Having given their informed, written consent

Exclusion Criteria:

* Contraindication to Electroconvulsive therapy (ECT), repeated Transcranial Magnetic Stimulation (rTMS), Magnetic Resonance Imaging (MRI), anesthesia
* Patients who have received ECT in the last 6 months
* Patients suffering from poorly stabilized epilepsy, serious neurological or systemic disorders
* Patients with a serious substance use disorder (other than nicotine or caffeine) according to DSM-5 criteria
* Patients suffering from severe hearing problems
* Subjects already treated with an electrical or magnetic stimulation technique
* Women who do not have adequate contraception, pregnant or breastfeeding women
* Being deprived of liberty by an administrative or judicial decision
* Patients participating or having participated in an interventional clinical trial within 30 days before the inclusion visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Response rate after 10 ECT | Day 0 and Day 40
  the percentage of patients who achieved a reduction of 50% or more from their initial Hamilton Depression Scale score (HAMD-21 items)

SECONDARY OUTCOMES:
The relative improvement of depressive symptoms throughout the study (assessed by a clinician) | Day 0, Day 4, Day 19, Day 26, Day 40
  the relative variation of HAMD-21
The relative improvement of depressive symptoms throughout the study (self-reported) | Day 0, Day 4, Day 19, Day 26, Day 40
  Quick Inventory of Depressive Symptomatology
Adverse effects | Day 4, Day 19, Day 26, Day 40
  Assessment of adverse effects with the Udvalg for Kliniske Undersogelser (UKU) side effects rating scale adapted to rTMS (adapted UKU)
Subjective assessment of memory | Day 4, Day 19, Day 26, Day 40
  Scores and variations in memory assessed with the Squire Subjective Memory Questionnaire (SSMQ)
Subjective assessment of cognitive functioning | Day 4, Day 19, Day 26, Day 40
  Scores and variations in cognitive functioning assessed with the Cognitive Failures Questionnaire (CFQ)
Global cognitive functioning (objective) | Day 0 and Day 40
  Scores and variations assessed with the Mini Mental Status Examination
Verbal memory performances (objective) | Day 0 and Day 40
  Scores and variations assessed with the RL/RI-16 test
Attention (objective) | Day 0 and Day 40
  Scores and variations assessed the D2 test of attention
Visuospatial and constructional ability (objective) | Day 0 and Day 40
  Scores and variations assessed with the Rey-Osterrieth complex figure test
Autobiographical memory (objective) | Day 0 and Day 40
  Scores and variations assessed with the autobiographical memory test (TEMPau)
Seizure threshold | Day 5, Day 9, Day 11, Day 16, Day 18, Day 23, Day 25, Day 30, Day 32, Day 37
  Seizure threshold during ECT
Seizure duration | Day 5, Day 9, Day 11, Day 16, Day 18, Day 23, Day 25, Day 30, Day 32, Day 37
  Seizure duration during ECT
Postictal Suppression | Day 5, Day 9, Day 11, Day 16, Day 18, Day 23, Day 25, Day 30, Day 32, Day 37
  Postictal Suppression during ECT
Dose of medication | Day 5, Day 9, Day 11, Day 16, Day 18, Day 23, Day 25, Day 30, Day 32, Day 37
  Dose of medication during ECT
Changes in regional gray matter density | Day 0 and Day 40
  Changes in regional gray matter density measured with 3D MRI
Changes in cortical thickness | Day 0 and Day 40
  Changes in cortical thickness measured with 3D MRI
Brain activity and biochemical changes | Day 0 and Day 40
  Changes measured with Resting state functional MRI and spectroscopy MRI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clabeau L, Moulier V, Kaczmarek B, Dalmont M, Batail JM, Bouaziz N, Brunelin J, Calvet B, Daudet C, Dollfus S, Domenech P, Drapier D, Galvao F, Gohier B, Harika-Germaneau G, Holtzmann J, Jaafari N, Jalenques I, Januel D, Kazour F, Laurin A, Letourneur F, Pouchon A, Samalin L, Sauvaget A, Szekely D, Vinckier F, Le Clezio C, Compere V, Gerardin E, Guillin O, Quesada P, Rotharmel M. A prospective multicentre double-blind randomized controlled trial evaluating clinical, cognitive and neural effects of potentiation of electroconvulsive therapy by repetitive transcranial magnetic stimulation in patients with treatment-resistant depression (STIMAGNECT 2). Trials. 2026 Jan 26. doi: 10.1186/s13063-025-09406-4. Online ahead of print. PMID 41582128